CLINICAL TRIAL: NCT03138109
Title: Analysis of Incidence and Risk Factors of Severe Cardiovascular Events in Patients With Diastolic Dysfunction
Status: Completed | Type: Observational
Sponsor: Yan Zhou, MD (Other)
Responsible Party: Sponsor-Investigator, Yan Zhou, MD, doctor, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: MACEDD
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Diastolic Dysfunction
Keywords: non-cardiac surgery; major adverse cardiac event

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- grade1&2 diastolic dysfunction: lower diastolic dysfunction exposure
- grade 3 diastolic dysfunction: higher diastolic dysfunction exposure

SUMMARY:
This retrospective cohort study was intended to analyze the incidence and risk factors of perioperative severe cardiovascular events in patients with diastolic dysfunction.

DETAILED DESCRIPTION:
The investigators retrospected patients underwent noncardiac surgery with pre-operative echocardiography and was diagnosed with diastolic dysfunction in 2015 in Peking University First Hospital. Patients' perioperative data were collected. Major adverse cardiovascular events(MACE), other complication incidence, and post-operative hospital stay were reviewed. propotional harzad ratio cox survival model was established. Risk and protective factors relative to MACE were analysed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older, with echocardiographic diagnosis of left ventricular diastolic dysfunction (while ejection fraction was > = 50%) conducted by cardiologist within 90 days before surgery.

Exclusion Criteria:

* congenital heart disease, moderate to severe valvular disease (stenosis or insufficiency), atrial fibrillation / atrial flutter, pericarditis, unsatisfied cardiac ultrasound image, ejection fraction < 50%, ASA greater than 4, or Echocardiography is missing or incomplete.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diastolic dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 4347 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
MACE | 30 days
  major cardiac complications

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhou, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- First hospital Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagueh SF, Appleton CP, Gillebert TC, Marino PN, Oh JK, Smiseth OA, Waggoner AD, Flachskampf FA, Pellikka PA, Evangelisa A. Recommendations for the evaluation of left ventricular diastolic function by echocardiography. Eur J Echocardiogr. 2009 Mar;10(2):165-93. doi: 10.1093/ejechocard/jep007. No abstract available. PMID 19270053
- [Background] Fischer M, Baessler A, Hense HW, Hengstenberg C, Muscholl M, Holmer S, Doring A, Broeckel U, Riegger G, Schunkert H. Prevalence of left ventricular diastolic dysfunction in the community. Results from a Doppler echocardiographic-based survey of a population sample. Eur Heart J. 2003 Feb;24(4):320-8. doi: 10.1016/s0195-668x(02)00428-1. PMID 12581679
- [Background] Roongsritong C, Qaddour A, Cox SL, Labib S, Bradley CA. Brain natriuretic peptide and diastolic dysfunction in the elderly: influence of gender. Congest Heart Fail. 2005 Mar-Apr;11(2):65-7. doi: 10.1111/j.1527-5299.2005.03747.x. PMID 15860970
- [Background] Redfield MM, Jacobsen SJ, Burnett JC Jr, Mahoney DW, Bailey KR, Rodeheffer RJ. Burden of systolic and diastolic ventricular dysfunction in the community: appreciating the scope of the heart failure epidemic. JAMA. 2003 Jan 8;289(2):194-202. doi: 10.1001/jama.289.2.194. PMID 12517230
- [Background] Fayad A, Ansari MT, Yang H, Ruddy T, Wells GA. Perioperative Diastolic Dysfunction in Patients Undergoing Noncardiac Surgery Is an Independent Risk Factor for Cardiovascular Events: A Systematic Review and Meta-analysis. Anesthesiology. 2016 Jul;125(1):72-91. doi: 10.1097/ALN.0000000000001132. PMID 27077638
- [Background] Devereaux PJ, Goldman L, Yusuf S, Gilbert K, Leslie K, Guyatt GH. Surveillance and prevention of major perioperative ischemic cardiac events in patients undergoing noncardiac surgery: a review. CMAJ. 2005 Sep 27;173(7):779-88. doi: 10.1503/cmaj.050316. PMID 16186585